CLINICAL TRIAL: NCT01935752
Title: Pathophysiological Mechanisms of Fibromuscular Dysplasia
Acronym: MeDyA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation pour la Recherche Médicale (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: P110301
Record Dates: First submitted 2013-09-02; First posted 2013-09-05 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Fibromuscular Dysplasia
Keywords: fibromuscular; dysplasia; endothelium; microparticles; microRNA
MeSH Terms: conditions — Fibromuscular Dysplasia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fibromuscular dysplasia (Other): Fibromuscular dysplasia:blood samples & vascular echotracking
  Interventions: Other: blood samples; Other: vascular echotracking
- healthy volunteer (Other): healthy volunteer:blood samples & vascular echotracking
  Interventions: Other: blood samples; Other: vascular echotracking
- hypertensive patients (Other): hypertensive patients:blood samples & vascular echotracking
  Interventions: Other: blood samples; Other: vascular echotracking

INTERVENTIONS:
Other: blood samples — blood samples
Other: vascular echotracking — endothelial function study and virtual histology study

SUMMARY:
Fibromuscular dysplasia is an non inflammatory non atherosclerotic obstructive arterial disease affecting mid-size arteries. It is considered as a rare vascular disease of unknown origin. Fibromuscular dysplasia may become symptomatic depending on location and severity of narrowing of the arterial lumen. for example,when a stenosis develops within a renal artery, arterial hypertension may develop. The cause of fibromuscular dysplasia is unknown. Several factors have been suggested to be associated with it: tobacco abuse or oestrogens. In order to progress into identifying possible causative mechanisms of the disease, we design a pathophysiology study destined to assess endothelial function in patients with fibromuscular dysplasia and to identify possible plasmatic biomarkers of the disease.

ELIGIBILITY:
Inclusion Criteria for patients with multifocal fibromuscular dysplasia:

* confirmed multifocal fibromuscular dysplasia
* diagnosed for less than 10 years
* without significant atherosclerotic disease or recent cardiovascular event
* Statins and antiplatelet drugs are forbidden
* hypertensive patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Comparison of circulating microparticles of patients vs. fibromuscular dysplasia with age and sex matched healthy volunteers and hypertensive patients | Once within 15 days

SECONDARY OUTCOMES:
Comparison of circulating micro RNAs (miR-143 ; miR-145) between the 3 arms | Once within 15 days
Comparison of matrixmetalloproteases between the 3 arms | Once within 15 days
Comparison of c-reactive protein between the 3 arms | Once within 15 days
Comparison of PLA2 between the 3 arms | Once within 15 days
Comparison of endothelium dependant vasodilation between the 3 arms | Once within 15 days
Comparison of endothelium independent vasodilation between the 3 arms | Once within 15 days
Comparison of pulse wave velocity between the 3 arms | Once within 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Michel Azizi, MD, PhD., Principal Investigator — HEGP, APHP, Paris, France
Locations (1):
- Cic9201, Hegp, Aphp,, Paris, France

REFERENCES:
- [Derived] Bruno RM, Marais L, Khettab H, Lorthioir A, Frank M, Jeunemaitre X, Laurent S, Boutouyrie P, Azizi M. Deep Vascular Phenotyping in Patients With Renal Multifocal Fibromuscular Dysplasia. Hypertension. 2019 Feb;73(2):371-378. doi: 10.1161/HYPERTENSIONAHA.118.12189. PMID 30624987